CLINICAL TRIAL: NCT03297827
Title: A Prospective Cytokine Registry Database of Stroke (Ischemic and Hemorrhagic) Patients.
Brief Title: Cytokine Registry Database of Stroke Patients
Acronym: CRISP
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: 17-315
Record Dates: First submitted 2017-09-21; First posted 2017-09-29 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2020-11

CONDITIONS: Acute Stroke; Acute Ischemic Stroke; Ischemic Stroke; Hemorrhagic Stroke
Keywords: diagnosis; inflammatory biomarkers; cytokines; interleukin; interferons
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood Specimens Urine Specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with stroke: Adult stroke patients with the stroke diagnosis will be recruited on admission to the University of New Mexico Hospital. Serum and Urine measurement of cytokines from two sets of serum and urine samples will be done on the admission and at the 24-hour mark respectively, form the specimens collected for the clinical purposes and are meant to be discarded. Consent will be taken from the patients to use these samples for our study.
  Interventions: Other: Serum and Urine measurement of cytokines.
- Patients without stroke: Age/Sex matched adult control patients without the diagnosis of stroke, myocardial infarction, inflammatory flare, acute trauma, neurodegenerative or neuroinflammatory disease (AD, PD, TM, PSP, etc.) except MS will be recruited on admission to the University of New Mexico Hospital. Serum and Urine measurement of cytokines from two sets of serum and urine samples will be done on the admission and at the 24-hour mark respectively, form the specimens collected for the clinical purposes and are meant to be discarded. Consent will be taken from the patients to use these samples for our study.
  Interventions: Other: Serum and Urine measurement of cytokines.

INTERVENTIONS:
Other: Serum and Urine measurement of cytokines. — To evaluate serum cytokine levels and identifying serum inflammatory markers (serum interleukin-33, IL-37, IL-36, IL-4, IL-6, IL-10, IL-17, IL-23, IL-1, TNF, PDGF, VEGFM TNFa, ANNULIN, MMP-9, MMP-12, NFk-B levels plus metabolic products like MPO, etc and glial factors like GMF, SI000B, GM6001) in patients with acute ischemic & hemorrhagic stroke.

SUMMARY:
Various molecules (cytokines: interleukins, interferons and neural proteins) found in human and animal blood are reported to be elevated in acute stroke (Ischemic and hemorrhagic). Cytokines can be pro-inflammatory or anti-inflammatory. There are studies confirming level changes in serum of humans in the setting of several rheumatologic and cardiovascular diseases. As new molecular markers (cytokines and neural tissue markers) are established in scientific literature, stroke scientists are interested to evaluate the role of these in the pathophysiology of stroke. Investigators intend to study the role of these molecules in the development of stroke.

Acute stroke treatment has advanced considerably in the last 10 years with the establishment of comprehensive stroke centers and approval of neuro-interventional techniques. However, the molecular advancement in stroke pathogenesis has yet to reach a milestone in the world of stroke treatment. In our opinion, creating a database of acute stroke patients containing all pertinent medical demographics and clinical information along with the laboratory data, molecular levels of pertinent cytokines/neural factors from consenting patients, will help us define and delineate the most relevant molecules that are altered in acute stroke patients and can help us further improve us understanding of the role of these in acute stroke and thereby hopefully help in the improvement of our understanding and management of stroke. Moreover, analyzing the cytokines in stroke and ICH patients would help understand their role in the acute phase, which may become potential therapeutic adjuncts for tPA and endovascular thrombectomy.

DETAILED DESCRIPTION:
Stroke is the fifth cause of all-cause mortality in US http://www.cdc.gov/stroke/facts.htm . Early identification and treatment not only prevent mortality but also morbidity. Recent advancement in the imaging and diagnostic technique and novel therapeutic modalities has dramatically helped to downgrade stroke from the list of top mortality index in the last 3 years. However, studies determining factors which help predict stroke outcome are still underway and much work needs to be done in this direction. Many factors currently are used to predict stroke outcome with varying results, for e.g. NIHSS is a good predictor of stroke outcome at 3 months; however, we need better predictors, outcome scales or outcome measures which are easy, reliable and has better specificity and sensitivity.

There is also some correlation of clinical and biochemical predictors in subarachnoid, cerebral venous thrombosis including Hunt and Hess, SAH score, WFNS-SAH grading among others with variable predictive quality. (Rosen et al; Neurocritical Care; April 2005, Volume 2, Issue 2, pp 110- 118: Subarachnoid hemorrhage grading scales).

During the acute phase of focal cerebral ischemia, there is an elevation of thrombin activity and a decline in fibrinolytic activity. Moreover, the role of pro-inflammatory cytokines has been proven in the last few decades, as markers of inflammation have been closely studied in mice models; there are indications that elevated levels correlate with the extent of ischemic injury. Various interleukins were found to be elevated in most if not all patients with acute ischemic stroke. Correlation of hemostatic (procoagulant and fibrinolytic markers) with inflammatory markers is under discussion, with no confirmed common marker identified as of yet.

As new cytokines and tissue markers are established in scientific literature, stroke scientists are interested in evaluating the role of these markers in the pathophysiology of stroke. The role of glial cell markers has been of remarkable interest. Recently, an astrocyte marker S100B has shown association with infarct size, neurological outcome, and prognosis. Moreover, analyzing the cytokines in stroke and ICH patients would help understand their role in the acute phase, which may become potential therapeutic adjuncts for tpa and endovascular thrombectomy. In summary, inflammation in acute stroke is an area of interest in the recent years, with the theoretical benefit of aborting the inflammatory chain during acute stroke might be useful in limiting stroke-related brain damage or hemorrhagic transformation in acute stroke.

ELIGIBILITY:
Inclusion Criteria:

1. All stroke patients (hemorrhagic and ischemic) presenting within 24 hours of onset who consent to our study.
2. Adult Male/Female patients ages >18 years old
3. Patients whose standard stroke admission order sets are obtained for clinical care.
4. Patients with a history of MS may be included for future subanalysis.

Exclusion Criteria:

1. History of prior stroke or any other neurodegenerative or neuroinflammatory disease (AD, PD, TM, PSP, etc.) except MS.
2. Individuals ages <18 year
3. Pregnant women
4. Prisoners

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Two sets of serum samples will be obtained and analyzed; one upon admission to the hospital, and the 2nd, the next morning after overnight fasting. Both sets of blood draw are done for a clinical purpose, and any extra stored sample that is drawn and not used by pathology will be used for the study. Twenty-five percent of the total stroke patient serum samples will be matched by appropriate controls to confirm the level changes in stroke patients. ELISA-PCR assays will be performed on serum samples.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the cytokine levels at the 24-hour mark from the baseline levels done at the time of admission for acute stroke. | 24 Hours
  Investigators will assess the variations in the levels of cytokines and inflammatory biomarkers at the 24-hour mark from the baseline levels done at the time of admission for acute stroke. Their correlation with each other may enable investigators to identify and streamline their efforts on only a few cytokines, interleukins, glial factors or metabolic products proved to be altered in acute stroke patients.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Torbey, MD, MPH, Study Chair — University of New Mexico; Atif Zafar, MD, Principal Investigator — University of New Mexico; Asad Ikram, MD, Study Director — University of New Mexico; Mudassir Farooqui, MD, MPH, Study Director — University of New Mexico
Locations (1):
- Department of Neurology, University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zafar A, Farooqui M, Ikram A, Suriya S, Kempuraj D, Khan M, Tasneem N, Qaryouti D, Quadri S, Adams HP, Ortega-Gutierrez S, Leira E, Zaheer A. Cytokines, brain proteins, and growth factors in acute stroke patients: A pilot study. Surg Neurol Int. 2021 Jul 27;12:366. doi: 10.25259/SNI_569_2021. eCollection 2021. PMID 34513133
- [Derived] Farooqui M, Ikram A, Suriya S, Saleem S, Quadri SA, Robinson M, Ortega-Gutierrez S, Qeadan F, Leira E, Paul S, Zafar A. Cytokine Registry In Stroke Patients (CRISP): Protocol of a prospective observational study. Medicine (Baltimore). 2020 Jul 10;99(28):e20921. doi: 10.1097/MD.0000000000020921. PMID 32664088
- [Derived] Zafar A, Ikram A, Jillella DV, Kempuraj D, Khan MM, Bushnaq S, Adam H, Ortega-Gutierrez S, Quadri SA, Farooqui M, Zaheer A, Leira EC. Measurement of Elevated IL-37 Levels in Acute Ischemic Brain Injury: A Cross-sectional Pilot Study. Cureus. 2017 Oct 11;9(10):e1767. doi: 10.7759/cureus.1767. PMID 29234571
- See also: Cytokines, brain proteins, and growth factors in acute stroke patients: A pilot study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8422456/